CLINICAL TRIAL: NCT06804954
Title: Internet-based Transdiagnostic Cognitive Behavior Therapy and Care As Usual for Primary Care Patients with Mental Ill-health (RCT-2: Subsyndromal Mental Ill-health)
Brief Title: Transdiagnostic Online CBT Vs. Care As Usual for Primary Care Patients with Subsyndromal Mental Ill-health ( PRIMARITA-2 )
Acronym: PRIMARITA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Hedman, Professor, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANS SUB 2024-06008-01 RCT-2
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Mental Ill-health
Keywords: Primary Care; Transdiagnostic CBT; Online treatment; Subsyndromal mental ill-health
MeSH Terms: interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online transdiagnostic CBT (Experimental): Participants randomized to this arm will receive the intervention online transdiagnostic CBT (see Interventions).
  Interventions: Behavioral: Online transdiagnostic CBT
- Primary care as usual (Active Comparator): Patients randomized to this study condition will receive health care services as usual in primary care.
  Interventions: Other: Primary care as usual

INTERVENTIONS:
Behavioral: Online transdiagnostic CBT — This treatment is provided through a secure web platform in which psychoeducation, worksheets, and exercises are presented in online modules similar to chapters in a book. Participants will receive weekly written feedback on their work and progress by a therapist who gives gradual access to the treatment modules. The lion's share of the contact between the therapist and the patient thus takes place through messages (similar to email) in the online treatment platform. It is however allowed to also have one to three face-to-face sessions on-site or through video calls to provide technical assistance and therapeutic support in accordance with the treatment model. Core components are: (a) psychoeducation about emotions and CBT, (b) functional analysis, (c) mindfulness practice, (d) breaking dysfunctional emotion-driven behaviors, and (e) exposure exercises.
  Arms: Online transdiagnostic CBT
Other: Primary care as usual — It is mandatory for primary care services in Stockholm, Sweden, to have staff with adequate competence in the assessment and treatment of common mental disorders. Typically, these patients are handled by general practitioners, psychologists, nurses, or social workers. As this comparator is intended to reflect real routine primary care, the interventions will not be controlled by the research project. We expect that participants allocated to this condition will receive an active treatment.
  Arms: Primary care as usual

SUMMARY:
The goal of this randomized controlled trial is to investigate if online transdiagnostic cognitive behavior therapy (CBT) can be effective in the treatment of subsyndromal mental ill-health in adult primary care patients. The main aim is to investigate:

if online transdiagnostic CBT yields superior symptomatic improvement compared to care-as-usual when given in a primary care context to patients with mental ill-health.

Researchers will compare online transdiagnostic CBT to primary care as usual to see if psychiatric symptoms can be reduced.

Participants will be randomized to online transdiagnostic CBT or primary care as usual. Participants in online transdiagnostic CBT will receive a cognitive behavioral treatment provided through a secure web platform in which psychoeducation, worksheets, and exercises are presented in online modules similar to chapters in a book. Participants will receive weekly written feedback on their work and progress by a therapist who gives gradual access to the treatment modules. The lion's share of the contact between the therapist and the patient thus takes place through messages (similar to email) in the online treatment platform.

Participants randomized to care as usual will receive health care services as usual in primary care. As this comparator is intended to reflect real routine primary care, the interventions will not be controlled by the research project, but the investigators expect that participants will receive an active treatment.

DETAILED DESCRIPTION:
Background: A large proportion of primary care patients with mental ill-health do not meet criteria for a manifest specific psychiatric disorder, but have subsyndromal mental ill-health that nonetheless requires treatment. The available research litterature regarding how to treat this patient group is scarce and the high demand for therapeutic services in primary care typically leads to low treatment accessibility. One possible and practical therapeutic solution is online transdiagnostic CBT, which draws on shared underlying mechanisms and is resource-efficient. There is still clear limitations in its evidence-base there is little data on how this method compares to primary care as usual for this patient group.

Purpose and aims: The overall purpose of the current trial is to build evidence for an accessible online transdiagnostic CBT for primary care patients with subsyndromal mental-ill health. A randomized controlled trial will be conducted where adult primary care patients with mental ill-health (but without manifest specific psychiatric disorder) will receive online transdiagnostic CBT or care as usual.

The main aim (I) of the study is to investigate if online transdiagnostic CBT yields superior symptomatic improvement compared to care-as-usual when given in a primary care context to patients with subsyndromal mental ill-health. Secondary aims are to investigate (II) if the treatment conditions are associated with improvement in quality of life, functional impairment, and neuroticism (III) moderators of treatment outcome, (IV) mediators of improvement, and (V) the cost-effectiveness (including effects on sickness absence) of online transdiagnostic CBT compared to primary care-as-usual. Should the trial fail to show a significant difference on the primary outcome, a secondary aim will also be to (VI) investigate if online transdiagnostic CBT is non-inferior to primary care as usual in reducing psychiatric symptoms.

Methods: This is a randomized controlled superiority trials where consecutively recruited adult primary care patients (N=500) are allocated in a 1:1 ratio to Internet-delivered transdiagnostic CBT or to primary care-as usual. This trial is part of larger project comprising two twin randomized controlled trials that are conducted in parallel where the difference between them is that the current trial will include patients with subsyndromal mental ill-health whereas the other (separately registered with clinicaltrials.gov) will include patients with a manifest psychiatric disorder.

Participants are consecutively recruited from the regular influx of primary care patients. Gustavsberg Primary Health Care Center in Region Stockholm, Sweden, is the basis, but additional primary care centers will be engaged to facilitate the recruitment and treatment of participants. The investigators expect that 10 to 20 primary care centers in Region Stockholm will be engaged for the recruitment and treatment of participants.

Patients who seek help for common mental health problems will be asked if they are interested in applying for the study. Those interested will undergo an assessment interview with a licensed clinician where all inclusion criteria are checked.

Measurements: See section Outcome Measures.

Treatment conditions: See section Arms and Interventions.

Data analysis: Change in the primary outcome measure will be analyzed using mixed effects linear regression. Fixed predictors in these analyses will be time, group and their interaction effect while taking individual variation in baseline symptom levels and change over time into account, i.e., random intercept and slope. Change from baseline to 10-week follow-up will be the primary endpoint. Power analyses show that to have 90% power to detect an effect size of d=0.25 (α=.05), given a correlation between measurements of 0.7, and an expected attrition of 15-20%, 250 participants will be needed in each arm (total sample size N=500). Should the main analysis show that there is a non-significant difference on the primary outcome, the investigators will conduct a secondary analysis of whether online transdiagnostic CBT is non-inferior to primary care-as-usual where the non-inferiority margin on the primary outcome is set to d=0.25, i.e., the bound of the one-sided 95% confidence interval must be within this margin for non-inferiority to be demonstrated. With 500 participants, 15-20% attrition, and a true null effect of zero, the study will have approximately 80% power to detect non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

To be included patients have to:

1. To be included patients have to: (a) have a subsyndromal mental health problem concerning anxiety, depressive symptoms, or stress-related ill-health that warrants treatment,
2. be at least 18 years old,
3. have regular access to a device with an Internet connection,
4. be able to read and write in Swedish,
5. have no severe psychiatric disorder that requires specialized psychiatric care, such as psychosis, bipolar disorder, or anorexia nervosa,
6. if on medication with monoamine agonist, have stable dosage in the past month,
7. have no on-going psychological treatment, and
8. provide written informed consent for participation and complete baseline assessment

Exclusion criteria:

As the targeted population in this trial is primary care patients with subsyndromal mental ill-health that do not have a manifest specific common mental disorder, patients will be excluded if they meet diagnostic criteria for an anxiety disorder (social phobia, panic disorder, agoraphobia, general anxiety disorder, or specific phobia), a health anxiety disorder (hypochondriasis or illness anxiety disorder), obsessive-compulsive disorder, depression (depression or dysthymia), or a stress-related disorder (exhaustion disorder, adjustment disorder, or post-traumatic stress disorder). Note that meeting diagnostic criteria for not otherwise specified disorders (e.g., anxiety not otherwise specified), mixed anxiety and depressive disorder, or disorders subsumed under "other" categories is not a reason for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2029-02-06 (Estimated); Study Completion 2029-02-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Depression Anxiety Stress Scales-21 (DASS-21) to 10-week, and 1-and 2- year follow-ups | Baseline, weeks 2, 4, 6, 8, 10 (primary endpoint), and 1-and 2-year follow-up
  This is a 21-item scale with a sum score range 0 to 126 where a higher score indicates more symptoms.

SECONDARY OUTCOMES:
Change in WHODAS from baseline to 10-week, and 1- and 2-year follow-ups | Baseline, week 10, 1- and 2-year follow-ups
  WHODAS is a 12-item measure of disability with a sum score range 0 to 100 where a higher score indicates more disability
Change in Work Ability Index from baseline to 10-week, and 1- and 2-year follow-ups | Baseline, week 10, 1- and 2-year follow-ups
  The Work Ability Index measures work ability with a sum score range 7 to 49 where a higher score indicates higher work ability
Change in Brunnsviken Brief Quality of Life Index from baseline to 10-week, and 1- and 2-year follow-ups | Baseline, week 10, 1- and 2-year follow-ups
  This is a measure of quality of life with a sum score range 0 to 96 where a higher score indicates higher quality of life
Change in sickness absence from 1 year before baseline to 1- and 2-year follow-ups | The 1-year period preceding baseline, 1- and 2-year periods after baseline
  Net days of sickness absence (including disability pension) will be calculated based on data from the Swedish Microdata for Analysis of Social Security (MiDAS) registry of the National Insurance Agency.
Change in EPQR-A Neuroticism scale from baseline to 10-week, and 1-and 2-year follow-ups | Baseline, week 10, 1- and 2-year follow-ups
  The EPQR-A (Eyesenck Personality Questionnaire Revised-Abbreviated) Neuroticism scale is a 6-item measure of neuroticism with a sum score range 0 to 6 where a higher score indicates more neuroticism.

OTHER OUTCOMES:
Client Satisfaction Questionnaire at 10-week follow-up | 10-week follow-up
  This is an 8-item measure of client satisfaction with the care received with a sum score range 8 to 32 where a higher score indicates higher client satisfaction
Negative Effects Questionnaire at 10-week follow-up | 10-week follow-up
  The Negative Effects Questionnaire is a 20-item measure of potential negative effects related to the received treatment. The participant marks (yes/no) if a negative effect has occurred from a list of common negative effects and rate to what extent this has affected the participant and to what extent it was related to treatment.
Credibility Scale (C-scale) 2 weeks after baseline | 2 weeks after baseline
  The C-scale is a measure of treatment credibility with a sum score range 0 to 50 where a higher score indicates higher treatment credibility
Change in EQ5D from baseline to 10-week, and 1- and 2-year follow-up | Baseline, week 10, 1- and 2-year follow-ups
  The EQ5D is a measure of health-related quality of life with a score range 0 to 1 where a higher score indicates higher quality of life. This measure will be used when calculating cost-utility in the health economic analysis.
Change in Difficulties in Emotion Regulation Scale-16 from baseline to 10-week, and 1- and 2-year follow-up follow-up | Baseline, weeks 2, 4, 6, 8, 10, and 1-and 2-year follow-up
  The Difficulties in Emotion Regulation Scale-16 is a scale with a sum score range 16 to 80 where a higher score indicates more difficulties in emotion regulation. This scale will be used as a putative mediator in mediation analysis.
Change in Brief Experiential Avoidance Questionnaire from baseline to 10-week, and 1- and 2-year follow-up | Baseline, weeks 2, 4, 6, 8, 10, and 1-and 2-year follow-up
  The Brief Experiential Avoidance Questionnaire is a scale with a sum score range 15 to 90 where a higher score indicates more experiential avoidance. This scale will be used as a putative mediator in mediation analysis.
Change in TIPI scale Openness to experience from baseline to 10-week follow-up, and 1- and 2-year follow-up | Baseline, weeks 2, 4, 6, 8, 10, and 1-and 2-year follow-up
  This is a subscale of the Ten Item Personality Inventory that measures the personality construct openness to experience with a sum score range 1 to 7 where a higher score indicates more openness to experience. This will be used as a statistical control mediator in mediation analysis, i.e., the investigators expect this scale will not mediate improvement.
Rate of healthcare consumption, by type | The 1-year period preceding baseline, 1- and 2-year periods after baseline
  Data will be collected from Region Stockholm's database (VAL) that provides information about all publicly healthcare provided in Stockholm County.
Socioeconomic information regarding income type | The 1-year period preceding baseline, 1- and 2-year periods after baseline
  Data will be retrieved from Statistics Sweden's LISA database (Longitudinal Integration Database for Health Insurance and Labour Market Studies) and include information about the type of income.
Number of participants with prescribed medication | The 1-year period preceding baseline, 1- and 2-year periods after baseline
  Registry data: National Board of Health and Welfares registry From the Prescribed Drug Register: Dispensed prescribed medications.
Clinical Global Impression Severity (CGI-S) at baseline | Baseline
  The CGI-S is a measure of global severity of psychiatric symptoms with a scale range 1 to 7 where a higher score indicates higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Hedman-Lagerlöf, PhD, professor, Principal Investigator — Region Stockholm and Karolinska Institutet
Locations (1):
- Region Stockholm, Gustavsberg Primary Care Center, Gustavsberg, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
The information collected in the study contains sensitive personal data and is protected by Swedish and European data secrecy regulations. Any data sharing is thus subject to assessment by relevant authorities and is not something the principal investigator can decide upon.